CLINICAL TRIAL: NCT00303862
Title: A Phase 2 Study of AZD2171 in Patients With Advanced Renal Cell Carcinoma
Brief Title: AZD2171 in Treating Patients With Refractory Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02686; NCI-2012-02686 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000460237; UCCRC-NCI-7111; NCI-7111; 14018A (Other: University of Chicago); 7111 (Other: CTEP); P30CA014599 (NIH); N01CM62201 (NIH); N01CM62209 (NIH)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2013-01

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cediranib

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive oral AZD2171 once daily for 4 weeks. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171; Recentin
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well AZD2171 works in treating patients with refractory metastatic kidney cancer. AZD2171 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with refractory metastatic renal cell carcinoma treated with AZD2171.

SECONDARY OBJECTIVES:

I. Determine the safety and tolerability of AZD2171 in these patients. II. Determine the feasibility of performing standardized delayed contrast-enhancement-MRI correlative studies across different institutions and platforms with data-sharing capability in patients with metastatic renal cell cancer.

III. Generate preliminary data regarding potential utility of pharmacogenomic and plasma/serum biomarkers of angiogenesis as predictive or prognostic markers for future investigations of AZD2171 and renal cell carcinoma.

OUTLINE: This is a multicenter study.

Patients receive oral AZD2171 once daily for 4 weeks. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed clear cell renal cell cancer

  * Must be predominantly metastatic disease
  * Refractory disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mmby conventional techniques or ≥ 10 mm by spiral CT scan
* No known brain metastases
* ECOG performance status 0-2
* Karnofsky 60-100%
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin normal
* Creatinine normal OR creatinine clearance > 60 mL/min
* Blood pressure < 140/90 mm Hg on 2 separate occasions not more than 6 weeks prior to enrollment and not less than 24 hours apart (stable antihypertensive regimen allowed)
* Mean QTc ≤ 470 msec (with Bazett's correction)
* Less than +1 proteinuria on two consecutive dipsticks taken no less than 1 week apart
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of familial long QT syndrome
* No cardiac arrhythmia
* No unstable angina pectoris
* No symptomatic congestive heart failure
* No New York Heart Association class III or IV disease
* No ongoing or active infection
* No hypertension
* No other uncontrolled intercurrent illness
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD2171
* No psychiatric illness or social situations that would limit compliance with study requirements
* See Disease Characteristics
* More than 4 weeks since prior radiotherapy and recovered
* More than 4 weeks since prior major surgery and recovered
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* More than 30 days since other prior investigational agents
* No prior therapy with vascular endothelial growth factor (VEGF) binding agents or VEGF receptor (VEGFR) tyrosine kinase inhibitors
* No more than 1 prior nonVEGF-directed systemic therapy for this disease
* No concurrent medication that may markedly affect renal function (e.g., vancomycin, amphotericin, ibuprofen, pentamidine)
* No combination antiretroviral therapy for HIV-positive patients
* No concurrent hematopoietic growth factors except epoetin alfa and bisphosphonates
* No concurrent hormones or other chemotherapeutic agents except for steroids given for adrenal failure and hormones administered for nondisease-related conditions (e.g. insulin for diabetes)
* No concurrent palliative or therapeutic radiation therapy
* No concurrent drugs or biologics with proarrhythmic potential
* No other concurrent investigational or commercial agents or therapies to treat the patient's malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between December, 2006 and July, 2007 at three institutions. The trial was terminated after 10 patients were enrolled due to insufficent accrual rate.
Period: Overall Study
Arm/Group | Treatment (Cediranib Maleate)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response
Description: Objective radiologic response as measured by RECIST criteria. (30% or greater shrinkage in the sum of the longest diameters of target lesions)
Time Frame: Up to 6 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 10
percentage of participants | 20 [2.5 to 55.6]

2. Secondary Outcome: Performance of DCE_MRI
Description: Binary (yes/no) indicator of whether a dynamic contrast-enhanced MRI (DCE-MRI)was successfully performed.
Time Frame: One month after initiating therapy
Population: Because trial was closed due to poor accrual, MRI data were not collected.
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 0

3. Secondary Outcome: KDR
Description: Kinase insert domain-containing vascular endothelial growth factor receptor
Time Frame: Day 28 after initiation of therapy
Population: Because trial was closed due to poor accrual, assays were not performed.
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 0

4. Secondary Outcome: eNOS
Description: Endothelial nitric oxide synthase gene (eNOS). Record genotype=number of minor alleles.
Time Frame: Baseline (prior to therapy)
Population: Because trial was closed due to poor accrual, assays were not performed.
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Grade 2 or higher
Arm/Group | Treatment (Cediranib Maleate)
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cediranib Maleate) (N=10)
Abdominal pain (Gastrointestinal disorders) | 2
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Anxiety (Psychiatric disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Ear, nose, and throat exam abnormal (Ear and labyrinth disorders) | 2
Fatigue (General disorders) | 4
Flatulence (Gastrointestinal disorders) | 1
GU bleeding (Reproductive system and breast disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Hand-and-foot syndrome (General disorders) | 5
Hyperglycemia (Endocrine disorders) | 1
Hypertension (Cardiac disorders) | 7
Hyperthyroidism (Endocrine disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypophophatemia (Metabolism and nutrition disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Infection (Infections and infestations) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Nausea/vomiting (Gastrointestinal disorders) | 1
Neurological disorder NOS (Nervous system disorders) | 1
Prostatic pain (General disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 3
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urogenital disorder (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less